CLINICAL TRIAL: NCT05764616
Title: Ultrasound Guided Parasternal Block Combined With Rectus Sheath Block for Cardiac Surgery Under Sternotomy: A Randomized Controlled Trial
Brief Title: Parasternal Block Combined With Rectus Sheath Block for Cardiac Surgery Under Sternotomy
Acronym: PARARECTUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Giuseppe Pascarella, Principal Investigator, Campus Bio-Medico University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PAR 06.23
Record Dates: First submitted 2023-02-27; First posted 2023-03-10 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Cardiac Disease; Surgery; Analgesia; Acute Pain; Postoperative Pain
MeSH Terms: conditions — Heart Diseases; Agnosia; Acute Pain; Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RECTUS group (Experimental): Patients will receive General Anesthesia combined with bilateral parasternal block and rectus sheath block
  Interventions: Procedure: PARASTERNAL BLOCK; Procedure: RECTUS SHEATH BLOCK
- CONTROL group (Active Comparator): Patients will receive General Anesthesia combined with bilateral parasternal block and infiltration of drainage exits sites with local anesthetic
  Interventions: Procedure: PARASTERNAL BLOCK; Procedure: LOCAL INFILTRATION OF DRAINAGE EXIT SITES

INTERVENTIONS:
Procedure: PARASTERNAL BLOCK — After induction of general anesthesia, an ultrasound-guided Parasternal Block will be performed with 20 mL of ropivacaine 0.5 % per side.
Procedure: LOCAL INFILTRATION OF DRAINAGE EXIT SITES — At the end of surgery, a local infiltration of drainage exit sites will be performed with 10 mL of ropivacaine 0.25% per side
  Arms: CONTROL group
Procedure: RECTUS SHEATH BLOCK — At the end of surgery, a rectus sheath block will be performed with 10 mL of ropivacaine 0.25% per side.
  Arms: RECTUS group

SUMMARY:
The aim of this randomized controlled trial is to examine the effect of ultrasound guided bilateral Parasternal Nerve Block combined with rectus sheath block on preoperative analgesia, opioid consumption and respiratory function in patients undergoing cardiac surgery via sternotomy. Half of participants will receive General Anesthesia combined with bilateral parasternal block and rectus sheath block while the other half receive General Anesthesia combined with bilateral parasternal block and infiltration of drainage exits sites with local anesthetic (without performing rectus sheath block)

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective cardiac surgery under median sternotomy
* Age >= 18 years
* American Society of Anesthesiologists (ASA) Status I-IV
* Approval and sign of the informed consent

Exclusion Criteria:

* Allergy to local anesthetics
* Puncture site infection
* Lack of signing of informed consent
* Age <18 years
* Emergency surgery
* ASA > IV
* preoperative acute respiratory failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2023-03-21 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2023-11-10 (Actual)

PRIMARY OUTCOMES:
Static Pain Score | 24 hours
  A numerical rating scale (NRS) from 0 (no pain) to 10 (worst imaginable pain) will be used to evaluate pain at rest during 24 hours after surgery
Dynamic Pain Score | 24 hours
  A numerical rating scale (NRS) from 0 (no pain) to 10 (worst imaginable pain) during movement will be used to evaluate pain at rest during 24 hours after surgery

SECONDARY OUTCOMES:
Intraoperative Fentanyl Consumption | 4 hours
  Total intravenous fentanyl administration (expressed in milligrams) during surgery
Morphine Consumption | 24 hours
  Total of intravenous morphine (expressed in milligrams) administered during the first 24 hours after surgery
Time of Extubation | 48 hours
  Interval between the end of surgery and patient's extubation
Respiratory performance at incentive spirometry | 48 hours
  Respiratory performance is assessed preoperatively and postoperatively (at extubation) by the number of balls raised during inspiration with the TRI-FLOW spirometer
Intensive Care Unit (ICU) Discharge Time | 120 hours
  Interval between patient arrival in ICU and discharge from ICU
Hospitalization Length of Stay | 30 days
  Total Hospital length of Stay (expressed in days)
Incidence of adverse events | 24 hours
  Any complications or side effects of the blocks, such as local infection, intravascular injection of local anesthetics and immediate systemic toxicity.
  Moreover, incidence of nausea, vomiting and postoperative respiratory complications will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Pascarella, MD, Principal Investigator — University Hospital Campus Biomedico of Rome
Locations (1):
- Campus Bio-medico University Hospital Foundation, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bloc S, Perot BP, Gibert H, Law Koune JD, Burg Y, Leclerc D, Vuitton AS, De La Jonquiere C, Luka M, Waldmann T, Vistarini N, Aubert S, Menager MM, Merzoug M, Naudin C, Squara P. Efficacy of parasternal block to decrease intraoperative opioid use in coronary artery bypass surgery via sternotomy: a randomized controlled trial. Reg Anesth Pain Med. 2021 Aug;46(8):671-678. doi: 10.1136/rapm-2020-102207. Epub 2021 May 14. PMID 33990437
- [Result] Barr AM, Tutungi E, Almeida AA. Parasternal intercostal block with ropivacaine for pain management after cardiac surgery: a double-blind, randomized, controlled trial. J Cardiothorac Vasc Anesth. 2007 Aug;21(4):547-53. doi: 10.1053/j.jvca.2006.09.003. Epub 2006 Dec 22. PMID 17678782
- [Result] Elbahrawy K, El-Deeb A. Rectus sheath block for postoperative analgesia in patients with mesenteric vascular occlusion undergoing laparotomy: A randomized single-blinded study. Anesth Essays Res. 2016 Sep-Dec;10(3):516-520. doi: 10.4103/0259-1162.179315. PMID 27746544
- [Result] Cibelli M, Brodier EA, Smith FG. Pectoralis-Intercostal-Rectus Sheath (PIRS) Plane Block With Catheters. A New Technique to Provide Analgesia in Cardiac Surgery. J Cardiothorac Vasc Anesth. 2020 Mar;34(3):846-847. doi: 10.1053/j.jvca.2019.09.014. Epub 2019 Sep 18. No abstract available. PMID 31590939
- [Result] Everett L, Davis TA, Deshpande SP, Mondal S. Implementation of Bilateral Rectus Sheath Blocks in Conjunction With Transversus Thoracis Plane and Pectointercostal Fascial Blocks for Immediate Postoperative Analgesia After Cardiac Surgery. Cureus. 2022 Jul 5;14(7):e26592. doi: 10.7759/cureus.26592. eCollection 2022 Jul. PMID 35936156
- [Derived] Strumia A, Pascarella G, Sarubbi D, Di Pumpo A, Costa F, Conti MC, Rizzo S, Stifano M, Mortini L, Cassibba A, Schiavoni L, Mattei A, Ruggiero A, Agro FE, Carassiti M, Cataldo R. Rectus sheath block added to parasternal block may improve postoperative pain control and respiratory performance after cardiac surgery: a superiority single-blinded randomized controlled clinical trial. Reg Anesth Pain Med. 2025 Sep 4;50(9):712-718. doi: 10.1136/rapm-2024-105430. PMID 38876800